CLINICAL TRIAL: NCT01866215
Title: Effects of Exercise on Fructose Metabolism
Acronym: FruEx2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University of Bern (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: University of Lausanne
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: gluconeogenesis; de novo lipogenesis; intramyocellular lipids; muscle glycogen; fructose
MeSH Terms: interventions — Exercise; Fructose; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Study1a (Experimental): exercice performed 90 min before 13C fructose meal ingestion
  Interventions: Other: exercise
- study 1b (Experimental): exercise performed 90 min after 13C fructose meal ingestion
  Interventions: Other: exercise
- study 1c (No Intervention): no exercise
- study 2a (Experimental): meals containing fructose, cream and whey proteins over 24 hours after a glycogen/intramyocellular lipid depleting exercise
  Interventions: Dietary Supplement: fructose
- study 2b (Active Comparator): meals containing glucose, cream and whey proteins over 24 hours after a glycogen/intramyocellular lipid depleting exercise
  Interventions: Dietary Supplement: glucose

INTERVENTIONS:
Other: exercise — cycling at 100W during 60 min
  Arms: Study1a; study 1b
Dietary Supplement: fructose — isocaloric nutrition with fructose, cream and whey protein during the 24 hour following a glycogen/intramyocellular lipid depleting exercise
  Arms: study 2a
Dietary Supplement: glucose — isocaloric nutrition with glucose, cream and whey protein during the 24 hour following a glycogen/intramyocellular lipid depleting exercise
  Arms: study 2b

SUMMARY:
A high fructose diet increases fasting and post-prandial triglyceride (TG) concentrations in sedentary healthy human subjects.These effects may be secondary to fructose-induced hepatic de novo lipogenesis. Recent evidence indicate that exercise can prevent fructose induced dyslipidemia.This study will evaluate

1. how exercise effects the metabolic fate of oral fructose 1a) when exercise is performed before fructose ingestion 1b) when exercise is performed after fructose ingestion Metabolic effects of exercise will be assessed in healthy male subjects by measuring fructose oxidation (13CO2 production), fructose conversion into glucose (13C glucose concentrations in blood) and hepatic fructose conversion into lipid (13C palmitate-very low density lipoprotein (VLDL) concentrations in blood) after ingestion of 13C-labelled fructose meals
2. how fructose and protein modulate muscle glycogen and intramyocellular lipid repletion after exercise Healthy male subjects will be fed various fructose, glucose, lipid and whey protein meals after a glycogen/intramyocellular lipid depleting exercise. The effects of meals' composition will be assessed after 24 hours by measuring intramyocellular lipids and glycogen using proton-magnetic resonance spectroscopy (MRS).

ELIGIBILITY:
Inclusion Criteria:

* males
* 18-40 years old
* 19 kg/m2>BMI>25kg/m2
* moderate to high usual physical activity
* non-smokers

Exclusion Criteria:

* family history of diabetes mellitus
* ECG anomaly
* any medication
* participation to blood spending or other clinical study in the 3 months before the beginning of this study
* consumption of drugs
* consumption of more than 50g alcool/week
* family history of food intolerance

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Plasma triglyceride | measurements in fasting conditions and every hour from 7:00 am to 4:00 pm (up to 9 hours)
  measurement of total and VLDL-TG concentrations in study 1
intramyocellular lipids | after glycogen/intramyocellular lipid depleting exercise and after 24 hour controlled feeding post exercise
  Measurement by 1H-MRS in muscle vastus lateralis in study 2
Fructose conversion into lipids | measured from 7:00 am to 4:00 pm in study 1 (up to 9 hours)
  Estimated from 13C palmitate-VLDL concentration

SECONDARY OUTCOMES:
Fructose conversion into glucose | measured between 7:00 am and 4:oo pm (up to 9 hours)
  measurements obtained from plasma 13C glucose concentrations and whole body glucose production measured by 6,6 d2 glucose in study 1)
intramyocellular glycogen concentrations | after glycogen/intramyocellular lipid depleting exercise and after 24 hour controlled feeding post exercise
  Measured by 1H-MRS in muscle vastus lateralis in study 2
fructose oxidation | measured from 7:00 am to 4:00 pm in study 1 (up to 9 hours)
  Calculated from breath 13CO2 production
exogenous lipid oxidation | measured from 7:00 am to 4:00 pm in study 2 (up to 9 hours)
  Lipids ingested will be labeled with 13C-triolein, and exogenous lipid oxidation will be measured from breath 13CO2 production

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Rosset R, Lecoultre V, Egli L, Cros J, Dokumaci AS, Zwygart K, Boesch C, Kreis R, Schneiter P, Tappy L. Postexercise repletion of muscle energy stores with fructose or glucose in mixed meals. Am J Clin Nutr. 2017 Mar;105(3):609-617. doi: 10.3945/ajcn.116.138214. Epub 2017 Jan 18. PMID 28100512
- [Derived] Egli L, Lecoultre V, Cros J, Rosset R, Marques AS, Schneiter P, Hodson L, Gabert L, Laville M, Tappy L. Exercise performed immediately after fructose ingestion enhances fructose oxidation and suppresses fructose storage. Am J Clin Nutr. 2016 Feb;103(2):348-55. doi: 10.3945/ajcn.115.116988. Epub 2015 Dec 23. PMID 26702120